CLINICAL TRIAL: NCT02897895
Title: Study to Evaluate the Value of the Follow-up of CALCIneurin Activity to MOdulate Calcineurin Inhibitors-induced Immunosuppression in Lung Transplantation
Acronym: CalciMo-TP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-16
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Lung Diseases
Keywords: Lung transplantation in end-stage lung diseases
MeSH Terms: conditions — Lung Diseases | interventions — Calcineurin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- new strategy of immunosuppression monitoring (Experimental): evaluation of calcineurin activity (CN-a) in combination with CNI blood levels
  Interventions: Biological: levels of CNI in whole blood; Biological: Calcineurin activity (CN-a) in peripheral blood mononuclear cells (PBMCs)
- strategy of reference (Active Comparator): CNI (inhibitor of Calcineurin) blood levels alone
  Interventions: Biological: levels of CNI in whole blood

INTERVENTIONS:
Biological: levels of CNI in whole blood
Biological: Calcineurin activity (CN-a) in peripheral blood mononuclear cells (PBMCs)
  Arms: new strategy of immunosuppression monitoring

SUMMARY:
The study is an interventional, multicentre, prospective, randomized, controlled, single-blind, comparative trial of two processes for adjusting the inhibitor of calcineurin (CNI) dosage in lung transplant recipients. Recipients will be stratified by transplant center and according to the underlying lung disease (affected with cystic fibrosis or not) and will be randomized to either evaluation of calcineurin activity (CN-a) in combination with CNI blood levels versus CNI blood levels alone in a 1:1 ratio. The objective is to compare the proportion of acute rejection that has required a specific curative treatment at 6 months after transplantation between patients in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient placed on the national waiting list for lung transplantation
* First de novo lung transplantation (single or double LTx)
* Prevention of allograft rejection by a usual immunosuppressive regimen including CNI (cyclosporine or tacrolimus)

Exclusion Criteria:

* Previous lung transplantation or other solid organ transplantation
* Combined lung transplantation with either liver or renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
number of episodes of acute rejection after LTx | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, Marseille, France